CLINICAL TRIAL: NCT05339139
Title: An Open-label, Prospective, Multicenter Study to Assess the SAfety of Regional Citrate Anticoagulation Delivered by the multiFiltratePRO System in Adult Patients Requiring Continuous Renal Replacement Therapy (SARCA Study)
Brief Title: SAfety of Regional Citrate Anticoagulation (SARCA Study)
Acronym: SARCA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ci-Ca-001
Record Dates: First submitted 2022-04-08; First posted 2022-04-21 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury; ESRD
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic | interventions — Dialysis

STUDY DESIGN:
Intervention Model Description: This is an open label, prospective, single-arm, multicenter study with adult patients requiring CRRT. In this study, the subjects will receive CRRT on the mFTPRO system with RCA.
  RCA treatment should be used until the end of CRRT. The circuit needs to be replaced after 72 hours of running time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Ci-Ca Arm (Experimental): The study population will include critically ill subjects who are a minimum of 18 years old, in an acute setting, requiring CRRT. the Subjects will receive Regional Citrate Anticoagulation (RCA) which will be delivered by MultiFiltiratePRO system
  Interventions: Combination Product: Dialysis

INTERVENTIONS:
Combination Product: Dialysis — In this study critically ill adult patients requiring Continuous Renal Replacement Therapy (CRRT) will receive Regional Citrate Anticoagulation (CRA) which will be delivered by multiFiltratePRO system.

SUMMARY:
This is an Open-label, Prospective, Multicenter Study to Assess the SAfety of Regional Citrate Anticoagulation Delivered by the multiFiltratePRO system in Adult Patients Requiring Continuous Renal Replacement Therapy (SARCA Study).

DETAILED DESCRIPTION:
In short, AKI is a major complication in intensive care patients, often occurring in the context of multiple organ failure, and some of these patients may need CRRT. The major advantage of CRRT is improved hemodynamic stability compared to intermittent HD. Continuous anticoagulation during CRRT may be needed to prevent premature clotting of the circuit and deliver the prescribed dialysis dose. Unfractionated heparin is the most commonly used anticoagulation during CRRT mainly as a result of familiarity, low cost, and ease of administration. But the main drawback is the risk of bleeding.

An alternative technique to avoid systemic anticoagulation is regional extracorporeal anticoagulation with citrate (RCA). The advantages of RCA are improved circuit patency and fewer bleeding complications. The use of RCA may also reduce the ICU staff workload. Studies have shown longer filter running times which reduced circuit change and set-up time. In addition, anticoagulation related bleeding, and CRRT-related blood transfusions were minimized. Therefore, CRRT with RCA might be more economical than conventional anticoagulation.

The study is to explore the possibility of using the multiFiltrate PRO system with the Ci-Ca module, Cifoban® (Trisodium citrate 4%), Calrecia® (Calcium chloride dihydrate), Ci-Ca dialysate K2 and K4, AV1000 (disposable cassette), and multiBic solution in subjects who are critically ill and receiving CRRT in an acute setting.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form by

   * The subject or
   * A legally authorized representative (LAR), if the subject is unable to consent
2. Adult patients ≥ 18 years old
3. Diagnosis of AKI or End-Stage Kidney Disease (ESKD) requiring CRRT
4. Vascular access - Dialysis Catheter with size and location per institutional practice

Exclusion Criteria:

1. Metabolic alkalosis as defined by serum bicarbonate greater than 30 mmol/L and arterial pH greater than 7.55
2. A female who is pregnant or breast feeding
3. Severe liver disease defined as International Normalized Ratio (INR) greater than 2.0 and total bilirubin greater than 5 mg/dl, and both aspartate aminotransferase (AST) and alanine aminotransferase (ALT) greater than 3 times upper limit of normal
4. Subjects currently enrolled in or who have completed any other investigational drug or device study within last 30 days prior to signing informed consent
5. Previous participation in a similar or the same study.
6. Subjects already on continuous renal replacement therapy
7. Subjects with active COVID-19 infection
8. Subjects cannot tolerate citrate therapy defined as severe liver disease (see exclusion criteria #3), shock with muscle hypoperfusion and known hypersensitivity to citrate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms and systemic ionized calcium level | Up to 1 month
  Defined as a symptomatic episode of delirium, coma, nausea, vomiting, constipation, muscle weakness, hypertension, bradycardia, deemed attributable to hypercalcemia with a confirmed systemic ionized calcium > 1.5mmol/L.
Arterial pH measure and bicarbonate level | Up to 1 month
  Arterial pH > 7.55 and bicarbonate > 30 mmol/L in the absence of exogenous bicarbonate administered
Serum sodium (Na) level | Up to 1 month
  Serum sodium (Na) level > 150 mmol/L and > 5 mmol/L rise in systemic Na above the prescribed CRRT fluids. Na level in the absence of hypertonic intravenous Na infusion
Drop in hemoglobin (Hgb) | Up to 1 month
  Bleeding resulting in more than 2 g/dL drop in hemoglobin (Hgb) in 24-hour period or need for transfusion
Symptoms and systemic ionized calcium level | Up to 1 month
  defined as a symptomatic episode of tetany/spasms, seizures, deemed attributable to hypocalcemia and with a confirmed systemic iCa < 0.85 mmol/L.
Symptoms and total-to-ionized calcium ratio | Up to 1 month
  Patients with impaired citrate metabolism or citrate overdose can exhibit citrate accumulation. Symptomatic citrate accumulation presents with symptoms of tetany/spasms, seizures, systemic hypocoagulability, hypotension, or cardiac events; and should be confirmed with:
  1. A total-to-ionized calcium ratio > 2.5; OR
  2. A total-to-ionized calcium ratio greater than 2.25 together with one or more of the following criteria:
     1. an increase in calcium supplementation,
     2. decreasing systemic ionized calcium, and
     3. metabolic acidosis. When a clinical presentation is possibly associated with an abnormal concentration of systemic ionized calcium or an altered acid-base balance, the labs ({Calcium: systemic ionized calcium, post-filter ionized calcium and total calcium}, bicarbonate, sodium, potassium, magnesium, phosphate) should be checked immediately.

SECONDARY OUTCOMES:
Circuit life | The life of a circuit is 72 hrs and then it needs to be replaced . Subject participation is upto 1 month.
  Circuit life is defined by time to circuit replacement

OTHER OUTCOMES:
Adverse Events | through study completion, an average of 1 year
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Stauss-Grabo, PhD, Study Director — Fresenius Medical Care North America
Locations (10):
- United States (10):
  - John L. McClellan Memorial Veterans' Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - Advent Health Orlando, Orlando, Florida
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University - Hospital, St Louis, Missouri
  - Intermountain Health, Murray, Utah